CLINICAL TRIAL: NCT04662450
Title: Evaluation and Management of Parturients' Pain Intensity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients.
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Jie Zhou, Assistant Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017P001416
Record Dates: First submitted 2018-07-31; First posted 2020-12-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Affective pain stimuli group (Experimental): affective/neutral word pairs
  Interventions: Behavioral: ABM affective pain stimuli
- Sensory pain stimuli group (Experimental): sensory/neutral word pairs
  Interventions: Behavioral: ABM sensory pain stimuli
- Control group (Placebo Comparator): affective/neutral and sensory/neutral word pairs
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: ABM affective pain stimuli — Patients undergo ABM training to shift attention away from affective pain stimuli
  Arms: Affective pain stimuli group
Behavioral: ABM sensory pain stimuli — Patients undergo ABM training to shift attention away from sensory pain stimuli
  Arms: Sensory pain stimuli group
Behavioral: Placebo — Patients undergo ABM training to receive affective/neutral and sensory/neutral word pairs
  Arms: Control group

SUMMARY:
The primary objective of this study is to examine the effects of Attentional Bias Modification (ABM) on the labor pain in parturients. One-third of the participants will undergo ABM training away from affective pain stimuli. One-third of the participants will undergo ABM training away from sensory pain stimuli. The rest of participants will be the control group.

DETAILED DESCRIPTION:
In recent years, significant attention has been paid to the attentional bias in patients with chronic pain. Studies found that Attentional Bias Modification (ABM) could reduce the pain intensity in participants with chronic pain. The investigator's goal is to evaluate the effects of ABM on labor pain and patient satisfaction with the labor and delivery experience.

ELIGIBILITY:
Inclusion Criteria:

* Parturients who are at 36 weeks gestation (at time of starting the study)

Exclusion Criteria:

1. Any patient who refuses
2. Patients with impaired decision-making capacity
3. Patients who are blind or extremely visually impaired
4. Patients who cannot understand or read English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturients
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effects of Attentional Bias Modification (ABM) on labor pain | 4 weeks (starting from 36-week gestation)
  Change in pain threshold and labor pain as measured by Fear of Pain Questionnaire (FPQ), Brief Pain Inventory (BPI) and McGill Pain Questionnaire (MPQ) before and after the ABM training.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhou, MD, MS, MBA, Principal Investigator — Harvard Medical School (HMS and HSDM)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Todd J, Sharpe L, Colagiuri B. Attentional bias modification and pain: The role of sensory and affective stimuli. Behav Res Ther. 2016 Aug;83:53-61. doi: 10.1016/j.brat.2016.06.002. Epub 2016 Jun 15. PMID 27327608
- [Result] Schoth DE, Georgallis T, Liossi C. Attentional bias modification in people with chronic pain: a proof of concept study. Cogn Behav Ther. 2013;42(3):233-43. doi: 10.1080/16506073.2013.777105. Epub 2013 Jun 4. PMID 23731349
- [Result] Duschek S, Werner NS, Limbert N, Winkelmann A, Montoya P. Attentional bias toward negative information in patients with fibromyalgia syndrome. Pain Med. 2014 Apr;15(4):603-12. doi: 10.1111/pme.12360. Epub 2014 Jan 21. PMID 24447855